CLINICAL TRIAL: NCT06686641
Title: Incidence of Macular Edema in a Uveitis Population of 1500 Patients
Brief Title: Incidence of Macular Edema in a Uveitis Population
Status: Active, not recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Jørgensen Cehofski, Dr. Lasse J. Cehofski, Aalborg University Hospital
Other Study IDs: ML45555
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Macular Edema; Non-infectious Uveitis
Keywords: Epidemiology of uveitis; Incidence of macular edema in a uveitis population; Management of macular edema secondary to uveitis; Uveitis; Macular Edema; Non infectious uveitis; Non-infectious uveitis
MeSH Terms: conditions — Macular Edema; Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-infectious uveitis patients treated at a hospitals in the North Denmark Region
  Interventions: Drug: Local and systemical treatment

INTERVENTIONS:
Drug: Local and systemical treatment — Evaluating the management of the edema including topical/local treatment (dexamethasone and NSAID, periocular injections, and dexamethasone intravitreal implant) and systemic treatment (prednisolone, DMARD, and biological agents, for example TNF-alpha inhibitors and interleukin-6 inhibitors). Moreover, the duration of any treatment as well as numbers of injections or implants.

SUMMARY:
Macular edema from uveitis is a serious condition that can lead to vision loss. Uveitis is an inflammation inside the eye, and macular edema is when fluid builds up in the central part of the retina, called the macula, which is crucial for clear vision. This fluid buildup can blur vision, sometimes severely. Managing this condition can be challenging and may require several treatments to reduce the fluid and protect sight. While we know macular edema is a common cause of vision loss in uveitis, there's limited data on how often it affects people in Europe

ELIGIBILITY:
Inclusion Criteria:

* Hospital-admitted patients in the North Denmark Region with non-infectious uveitis.
* Both juvenile and adult patients.
* Diagnosed with non-infectious uveitis by a medical doctor.
* Patients presenting with unspecific macular edema may be included if medical records indicate uveitis as the cause of the edema.

Exclusion Criteria:

* Patients incorrectly classified as having uveitis based on their medical records (no confirmed diagnosis of uveitis).
* Patients with infectious uveitis.
* Macular edema due to other cause than uveitis will not count as uveitis associated edema

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of all uveitis patients treated at hospitals in the North Denmark Region.The included study population consists of all patients with a primary or secondary first-time discharge diagnosis of uveitis from the ophthalmologic department at Aalborg University Hospital in the North Denmark Region. Both inpatient and outpatient diagnoses are included. The following ICD-10 codes for uveitis will be included: DH200 acute and subacute anterior uveitis, DH201 Chronic anterior uveitis, DH209 anterior uveitis unspecified, DH208 other anterior uveitis, DH300 focal posterior uveitis, DH309 posterior uveitis unspecified, DH308 other posterior uveitis, DH301 disseminated posterior uveitis, DH302 intermediate uveitis, and DH441E panuveitis
Sampling Method: Non-Probability Sample
Enrollment: 1550 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Macular Edema in patients with Uveitis | 10 years
  The outcome of interest is macular edema in non-infectious uveitis. We will estimate the incidence rate and cumulative incidence of macular edema in patients with uveitis. In addition, the population will be stratified according to sex, age, non-infectious uveitis subtype, HLA- subtype, and ethnicity (if available), and the rate and risk of macular edema will be assessed for each strata. The incidence rate for macular edema will be calculated for a 1-10 years follow-up periods. Furthermore, the cumulative incidence will be assessed using the Aalen Johansen estimator. The stratified groups will be compared using a cox proportional hazard model to quantify the differences between the respective groups. Patients will be excluded if essential information is missing in their medical journal. Follow-up will terminate in case the patient moves to an address outside the North Denmark Region.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse J Cehofski, MD, P.h.d, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ørskov et al. J Pers Med. 2023 8;13(6):970
- [Background] Xue YQ, Xiao JA, Chen Y. Frequency and Treatment Regimens of Macular Edema in 1946 Consecutive Patients with Noninfectious Uveitis at a Tertiary Ophthalmic Center in Shaanxi, China. Ophthalmol Ther. 2023 Oct;12(5):2609-2619. doi: 10.1007/s40123-023-00763-4. Epub 2023 Jul 13. PMID 37440091
- [Background] Koronis S, Stavrakas P, Balidis M, Kozeis N, Tranos PG. Update in treatment of uveitic macular edema. Drug Des Devel Ther. 2019 Feb 19;13:667-680. doi: 10.2147/DDDT.S166092. eCollection 2019. PMID 30858697
- [Background] Massa H, Pipis SY, Adewoyin T, Vergados A, Patra S, Panos GD. Macular edema associated with non-infectious uveitis: pathophysiology, etiology, prevalence, impact and management challenges. Clin Ophthalmol. 2019 Sep 10;13:1761-1777. doi: 10.2147/OPTH.S180580. eCollection 2019. PMID 31571815